CLINICAL TRIAL: NCT04234984
Title: A Retrospective Single-center Cohort Study on Patients With Chronic Knee Pain Treated With Conventional Radiofrequency of the Genicular Nerves
Brief Title: Patients With Chronic Knee Pain Treated With Conventional Radiofrequency of the Genicular Nerves
Acronym: RECORGEN
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Jan Van Zundert, Principal Investigator, Ziekenhuis Oost-Limburg
Other Study IDs: RECORGEN
Record Dates: First submitted 2020-01-07; First posted 2020-01-21 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Chronic Knee Pain
Keywords: Conventional radiofrequency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conventional radiofrequency (RF) treatment: All patients with chronic knee pain who qualify for a conventional RF treatment of the genicular nerves

SUMMARY:
Management of chronic knee pain remains a challenge to the treating physician. A radiofrequency treatment of the genicular nerves is a not yet established but promising technique. This procedure is minimal invasive and has few adverse events. For these reasons it can be advantageous and fulfilling the unmet needs of these chronic knee pain patients warranting further research of its efficacy.

To investigate this efficacy, all patients treated with radiofrequency ablation in the multidisciplinary chronic pain center between 1 September 2017 and 31 December 2019 with exclusion of patients with chronic widespread pain, will be retrospectively analyzed in a single-center cohort.

DETAILED DESCRIPTION:
This project has as primary objective the evaluation of treatment success of a conventional radiofrequency treatment of the genicular nerves in patients diagnosed with chronic knee pain due to osteoarthritis of the knee or persistent post-surgical pain (PPSP) at six weeks post treatment. Secondary objectives are evaluation of treatment effect at a third time point at the end of the inclusion period, subgroup analysis of treatment success based on indication to treatment, evaluation of subjective functional improvement and change in analgesics, estimation of the duration of effect of the treatment and adverse events.

This study includes all patients treated with radiofrequency ablation in the multidisciplinary chronic pain center in Ziekenhuis Oost-Limburg, Campus Sint-Barbara between 1 September 2017 and 31 December 2019 with exclusion of patients with chronic widespread pain.

The main study outcome is the proportion of patients with a global perceived effect of at least 50% at 6 weeks post intervention. Secondary outcomes include reduction in pain intensity, measured by Numeric Rating Scale (NRS) at six weeks and at a third time point, global perceived effect at a third time point, subjective change in physical functioning, duration effect of the treatment, use of strong opioids, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic knee pain who qualify for a conventional RF treatment of the genicular nerves

Exclusion Criteria:

* A negative diagnostic block with lidocaine 2% 1 ml of the three genicular nerves defined as less than 50% pain reduction
* Chronic widespread pain

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with chronic knee pain who qualify for a conventional RF treatment of the genicular nerves can be possible candidated for this retrospective study
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-01-26 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Zundert, MD PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Derived] Belba A, Vanneste T, Van Kuijk SMJ, Mesotten D, Mestrum R, Van Boxem K, Van Lantschoot A, Bellemans J, Van de Velde M, Van Zundert J. A retrospective study on patients with chronic knee pain treated with ultrasound-guided radiofrequency of the genicular nerves (RECORGEN trial). Pain Pract. 2022 Mar;22(3):340-348. doi: 10.1111/papr.13088. Epub 2021 Nov 9. PMID 34716965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2017 to June 2020. Patients receiving treatment in Hospital Oost-Limburg, Genk, Belgium.
Pre-assignment Details: Excluded patients (n=7): Chronic widespread pain (n=7)
Groups:
- Conventional Radiofrequency (RF) Treatment: All patients with chronic knee pain who qualify for a conventional radiofrequency (RF) treatment of the genicular nerves
Period: Follow-up at 6 Weeks
Arm/Group | Conventional Radiofrequency (RF) Treatment
Started | 61
Completed | 59
Not Completed | 2
Not completed — Lost to Follow-up | 2
Period: Follow-up at the Second Time Point
Arm/Group | Conventional Radiofrequency (RF) Treatment
Started (All patients experiencing a successful treatment at 6 weeks were followed up at the second time point.) | 19
Completed | 17
Not Completed | 2
Not completed — Death | 1
Not completed — Mentally unable to fill in the questionnaire | 1

BASELINE CHARACTERISTICS:
Groups:
- Degenerative Knee Pain: All patients with chronic knee pain who suffer from osteoarthritis (OA), soft tissue (e.g., ligament) disease and posttraumatic pain.
- Persistent Post-surgical Pain (PPSP): All patients with chronic knee pain who suffer from PPSP after all types orthopaedic surgeries of the knee.
- Total: Total of all reporting groups
Arm/Group | Degenerative Knee Pain | Persistent Post-surgical Pain (PPSP) | Total
Number analyzed (Participants) | 13 | 46 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (15.9) | 66.9 (13.9) | 62.6 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 33 | 40
  Male | 6 | 13 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Index knee [Number; unit: participants]
  Right | 9 | 18 | 27
  Left | 4 | 28 | 32
Patients on strong opioids at baseline consultation [Count of Participants; unit: Participants]
  No use of strong opioids | 10 | 33 | 43
  Use of strong opioids | 3 | 13 | 16
Mean NRS (± SD) prior to RF treatment [Mean (Standard Deviation); unit: units on a scale.] — Mean Numerical Rating Scale (NRS) (± standard deviation (SD)) prior to Radiofrequency treatment The NRS score is a score form 0 to 10. Patients are asked to rate their pain from 0 to 10 where 0 mean ' No pain' while 10 means ' Worst pain'.
  units on a scale. | 7.8 (1.7) | 7.3 (1.7) | 7.4 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Reaching Treatment Succes at 6 Weeks Defined as Global Perceived Effect (GPE) of ≥ 50% Compared to Baseline.
Description: Treatment success is defined as a global perceived effect (GPE) of at least 50% at measurement time point compared to baseline.
  Global perceived effect (GPE) scales are used as an overall outcome measure for patients with pain, as they may cover additional aspects to pain relief and physical function that are important to the individual. Patients are asked to response on the question of how the treatment influenced the pain symptoms. The patients were asked to expres their answer in percentage where 0 % ( no improvement) to 100 (total improvement, the symptoms are gone).
Time Frame: 6 weeks after treatment
Measure: Count of Participants; unit: Participants
Groups:
- Degenerative Knee Pain: All patients with chronic knee pain who suffer from OA, soft tissue (e.g., ligament) disease and posttraumatic pain.
- PPSP: All patients with chronic knee pain who suffer from PPSP after all types orthopaedic surgeries of the knee.
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 13 | 46
Participants | 4 | 15

2. Secondary Outcome: The Number of Participants With NRS Reduction ≥50% Compared to Baseline
Description: The numeric rating scale (NRS) is used to assess pain intensity varying from 0 (no pain) to 10 (intense pain). This scale was retrieved retrospectively out of the patient file.
  NRS reduction ≥50% is calculated using the NRS at 6 weeks compared to the NRS at baseline.
Time Frame: 6 weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 13 | 46
Participants | 4 | 9

3. Secondary Outcome: The Patient's NRS
Description: The numeric rating scale (NRS) is used to assess pain intensity varying from 0 (no pain) to 10 (intense pain). This scale will be asked telephonically to the patient.
Time Frame: after retrieval of informed consent, ranging from 6 weeks to 2.5 years after the procedure
Population: At the second time point: 4 patients with degenerative knee pain and 13 patients with PPSP were analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 13 | 46
score on a scale
  Mean NRS at 6 weeks | 5.6 (1.9) | 7.3 (1.7)
  Mean NRS in treatment success group: number analyzed (Participants) | 4 | 15
  Mean NRS in treatment success group | 2.8 (1.5) | 3.4 (1.7)
  Mean NRS in treatment failure group: number analyzed (Participants) | 9 | 31
  Mean NRS in treatment failure group | 7.1 (2.4) | 7.5 (1.5)
  Mean NRS at the second time point: number analyzed (Participants) | 4 | 13
  Mean NRS at the second time point | 5.3 (2.0) | 5.5 (1.9)
  Mean NRS at the second time point in patients with GPE ≥50%: number analyzed (Participants) | 2 | 4
  Mean NRS at the second time point in patients with GPE ≥50% | 4.0 (0.0) | 3.8 (2.2)
  Mean NRS at the second time point in patients with GPE <50%: number analyzed (Participants) | 2 | 9
  Mean NRS at the second time point in patients with GPE <50% | 6.0 (2.0) | 6.6 (0.8)

4. Secondary Outcome: The Number of Patients With Subjective Increase in Physical Functioning at the Second Time Point
Description: The question 'Do you experience at the moment functional improvement in comparison with before the treatment?' is asked telephonically to the patient. The possible answers are 'no increase in physical functioning' and ' yes, there was an increase in physical funcitoning'. An increase in physical functioning is the best outcome.
Time Frame: after retrieval of informed consent, ranging from 6 weeks to 2.5 years after the procedure
Population: 19 patients in total reached treatment succes at 6 weeks, 4 of which suffered from degenerative knee pain and 13 from PPSP. Two of these patients were excluded from analysis due to death and being mentally unable to fulfill the questionnaire. As a result 17 patients were analyzed for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 4 | 13
Participants | 1 | 6

5. Secondary Outcome: The Number of Pariticipants Using Strong Opioids
Description: The change in use of strong opioids is retrieved retrospectively out of the patient file. The answer to the use of strong opioids is yes or no. No use of strong opioids is a better outcome.
Time Frame: 6 weeks after treatment
Population: Strong opioid use is measured firstly in both subgroups and secondly in the treatment success and treatment failure group.
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 13 | 46
Participants
  Patients on strong opioids | 3 | 8
  Patients on strong opioids in treatment success group: number analyzed (Participants) | 4 | 15
  Patients on strong opioids in treatment success group | 1 | 3
  Patients on strong opioids in treatment failure group: number analyzed (Participants) | 9 | 31
  Patients on strong opioids in treatment failure group | 2 | 5

6. Secondary Outcome: Strong Opioid Use at the Second Time Point
Description: The change in use of strong opioids is asked telephonically to the patient.
Time Frame: after retrieval of informed consent, ranging from 6 weeks to 2.5 years after the procedure
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 4 | 13
Participants | 1 | 5

7. Secondary Outcome: The Number of Participants Reaching Treatment Success After Retrieval of the Informed Consent Defined as GPE of ≥ 50% Compared to Baseline.
Description: as for outcome 1
Time Frame: after retrieval of informed consent, ranging from 6 weeks to 2.5 years after the procedure
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 4 | 13
Participants | 2 | 4

8. Secondary Outcome: Number of Participants With Post-treatment Complications
Description: Adverse events related to the conventional radiofrequency therapy will be assessed. This will be assessed retrospectively in the patient file according to the standard of care consultation at 6 weeks after treatment.
Time Frame: 6 weeks after treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 13 | 46
Participants
  Adverse events | 3 | 6
  Severe adverse events | 0 | 1

9. Secondary Outcome: Number of Participants With Post-treatment Complications
Description: Adverse events related to the conventional radiofrequency therapy will be assessed telephonically
Time Frame: after retrieval of informed consent, ranging from 6 weeks to 2.5 years after the procedure
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Knee Pain | PPSP
Number analyzed (Participants) | 4 | 13
Participants
  Adverse events | 0 | 1
  Severe adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Collection of data happened in a time period that was different for every patient varying from 6 weeks to 2.5 years
Description: Adverse events were defined as any undesirable experience occurring to a subject during the study that is related to the investigational intervention.
Arm/Group | Degenerative Knee Pain | PPSP
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/46
Other Adverse Events (participants affected / at risk) | 3/13 | 5/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degenerative Knee Pain (N=13) | PPSP (N=46)
Complex regional pain syndrome (CRPS) (Nervous system disorders) | 0 (0) | 1 (1) — CRPS of the treated knee
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degenerative Knee Pain (N=13) | PPSP (N=46)
Instability while walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Instability, no fall
Hypoesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Increase in pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Self-limiting hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cracking of the joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1. One of the limitations of this study is inherent to its retrospective nature.
2. A second limitation is that comparison with previous studies is difficult due to the use of ultrasound as guidance for the procedure as most of the studies use fluoroscopy-guided RF.
3. Another limitation concerns the subgroup analysis of degenerative knee pain. These results need to be interpreted with caution due to the small number of patients included in this group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04234984/Prot_SAP_000.pdf